CLINICAL TRIAL: NCT04959929
Title: Wearable Focal Vibration for Chemotherapy-Induced Peripheral Neuropathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12621
Record Dates: First submitted 2021-03-29; First posted 2021-07-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: focal vibration; wearable; in-home rehabilitation; chemotherapy-induced peripheral neuropathy; CIPN; lower extremity

STUDY DESIGN:
Intervention Model Description: All participants will be assigned to a single group that will receive focal vibration therapy using Myovolt.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Focal vibration therapy (Experimental): Myovolt delivers vibration with a frequency between 50-80 Hz. Myovolt intensity will be set to ~up to 2X the participant's initial Myovolt perception threshold. If the stimulation does not feel strong, the participant will be asked to manually increase the intensity until it feels strong but comfortable.
  Interventions: Device: Focal vibration therapy

INTERVENTIONS:
Device: Focal vibration therapy — Myovolt is a wearable rehabilitative device that delivers vibration to the region of the body where the motors are worn. Participants are asked to apply the vibration to specific leg locations twice a day, for about 30 minutes at a time, and to record their response using a provided log. They may be asked to try applying the device at different location or using different vibration parameters (pulse frequency or intensity).
  Other Names: Myovolt

SUMMARY:
This study will perform an early Phase I feasibility study with single-arm, double-baseline repeated measured design. The investigators will test the feasibility of using focal vibration to improve symptoms of persistent CIPN.

DETAILED DESCRIPTION:
This is an initial Phase I single-site, single-arm, double-baseline repeated measures feasibility study of wearable focal vibration (FV with Myovolt) for persistent chemotherapy-induced peripheral neuropathy. We will enroll up to 15 cancer survivors who are cancer-free and meet all other inclusion/ exclusion criteria, including CIPN symptoms at least 3 months after final chemotherapy infusion. Participants will undergo baseline assessments (V1) of questionnaires and performance tests, and may repeat these tests within a few days as a double-baseline (V2). In addition, they complete 7-days of baseline symptom monitoring by diary before starting 6 weeks of daily at-home therapy with a Myovolt wearable FV device. A study coach will check in by phone or video calls during the intervention period. Participants undergo post-testing immediately after the 6-week intervention (V3), and after another 6 weeks without FV (V4). In total, participants attend 3-4 onsite study visits, a 6-week intervention period with weekly remote check-in contact from the study team, and a 6-week intervention-free follow-up period with at least one remote check-in. Participants will keep a provided daily symptom diary during the primary study period (i.e., 6 weeks), and at least weekly in the 6-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Cancer patients with current symptoms of chemotherapy induced peripheral neuropathy affecting the feet, persisting for at least 3 months after completion of chemotherapy, and not substantially improving in recent weeks. The CIPN must be painful, or severe enough to interfere with function, activities, or participation (generally NCI-CTCAE Grade II)
* Clinically stable to participate in study assessments and the intervention (at a minimum, able to stand independently from a chair and walk household distances without help from another person)
* Able to read and speak English, give a voluntary written consent
* Sufficient cognition to consent, confirmed by recall of key study points
* Use of pain medications (opioids, anti-convulsants, and antidepressants) must be stable in the two weeks prior to study enrollment, and the participant must agree to avoid significant changes in pain medication regimen during the period of active study participation, and to notify the study team if medications change

Exclusion Criteria:

* Neuropathy (known or suspected) of any etiology other than chemotherapy or diabetes (for example, due to alcohol, vitamin deficiency, autoimmune disorder, CMT, idiopathic
* Unsafe/unable to self-apply the focal vibration intervention for any reason (for example, insufficient hand dexterity or cognitive executive function
* Recent or fluctuating musculoskeletal injury or lesion that would impact physical performance
* Lower limb deficiency/amputations
* Pregnant, or planning to get pregnant in the next 6 months. Pre-menopausal females who enroll agree to notify the study team as soon as possible should they become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of enrollment | Baseline
  Percent of interested individuals who enrolled.
Adherence to Myovolt focal vibration | After 6-week intervention
  Number of completed days and sessions of Number of days (or sessions) the intervention was worn, as a percentage of the number of days (or sessions) the device was prescribed.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity-12 (FACT-GOG/NTX-12) Symptom Inventory | Change from Baseline after 6-week Intervention
  The FACT-GOG/Ntx-12 is a composite measure of CIPN symptoms and functional impairments and related quality of life, scored from 0 to 48 where a higher score indicates worse neuropathy symptoms.
Neuropathy Total Symptom Score-6 (NTSS-6) | Change from Baseline after 6-week Intervention
  The NTSS-6 rates neuropathic symptoms (severity and frequency) in 6-categories. Scores range from 0 to 21.96, and higher scores indicate higher symptom burden.
Patient Neurotoxicity Questionnaire (PNQ) | Change from Baseline after 6-week Intervention
  The PNQ grades the extent of sensory and motor neuropathy in cancer cohorts scored from grade A (no neuropathy, also Grade 0) to grade E (severe neuropathy, also Grade 4) for both sensory and motor symptoms.
Global Rating of Change (GROC) scale | After 6-week withdrawal period
  The GROC scale is a universal clinical outcome providing a simple but comprehensive "umbrella" patient-perspective of change with scores ranging from -5 (very much worse) to 0 (unchanged) to +5 (completely recovered).
Long-term retention | After 6-week withdrawal period
  Number of enrolled individuals retained for long-term follow-up(after 6-week withdrawal period), and reasons for loss to follow-up, when available.
Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity-12 (FACT-GOG/NTX-12) Physical Well-Being Subscale | Change from Baseline after 6-week Intervention
  The FACT-GOG/Ntx-12 PWB subscale is a patient-report measure of physical symptoms and function. Scored from 0 to 28, higher scores indicate better well-being.
Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity-12 (FACT-GOG/NTX-12) Functional Well-Being Subscale | Change from Baseline after 6-week Intervention
  The FACT-GOG/Ntx-12 FWB subscale is a patient-report measure of functional well-being with questions about work, leisure and sleep, and a summary quality of life(QoL)rating. Scores range from 0 to 28, higher scores indicate better well-being and QoL.
Manual Muscle Testing (MMT) of Toes | Change from Baseline after 6-week Intervention
  MMT assesses muscle strength by an assessor applying pressure against the toes as the participant lifts or curls their toes and is rated from 0 (weakest) to 5 (strongest).
Toe Strength using a quantifiable toe measurement device | Change from Baseline after 6-week Intervention
  The toe strength quantifiable toe measurement device measures toe strength by reading force measurements when participants sit with foot strapped on a portable base of a load-cell prototype device of PI Dr. Hile and her team, with toe inserted into housing against which they pull up for a few seconds, or press down.
Vibration Perception Threshold using Biothesiometer | Change from Baseline after 6-week Intervention
  Vibratory threshold will be measured by a non-invasive vibrating probe (biothesiometer) placed on the skin. Vibration intensity is measured in frequency where the frequency is increased until the participant reports feeling it (eyes closed) from 0 to 50 Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hile, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Stephenson Cancer Center, OU Health, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data might be shared with permission from the funder and PI per request.
Supporting Information: Study Protocol, SAP
Time Frame: After study completion and publication of primary outcomes
Access Criteria: Only de-identified data will be shared with permission from the funder and PI per request

REFERENCES:
- [Background] Winters-Stone KM, Horak F, Jacobs PG, Trubowitz P, Dieckmann NF, Stoyles S, Faithfull S. Falls, Functioning, and Disability Among Women With Persistent Symptoms of Chemotherapy-Induced Peripheral Neuropathy. J Clin Oncol. 2017 Aug 10;35(23):2604-2612. doi: 10.1200/JCO.2016.71.3552. Epub 2017 Jun 6. PMID 28586243
- [Background] Monfort SM, Pan X, Patrick R, Ramaswamy B, Wesolowski R, Naughton MJ, Loprinzi CL, Chaudhari AMW, Lustberg MB. Gait, balance, and patient-reported outcomes during taxane-based chemotherapy in early-stage breast cancer patients. Breast Cancer Res Treat. 2017 Jul;164(1):69-77. doi: 10.1007/s10549-017-4230-8. Epub 2017 Apr 3. PMID 28374323
- [Background] Miaskowski C, Mastick J, Paul SM, Abrams G, Cheung S, Sabes JH, Kober KM, Schumacher M, Conley YP, Topp K, Smoot B, Mausisa G, Mazor M, Wallhagen M, Levine JD. Impact of chemotherapy-induced neurotoxicities on adult cancer survivors' symptom burden and quality of life. J Cancer Surviv. 2018 Apr;12(2):234-245. doi: 10.1007/s11764-017-0662-8. Epub 2017 Nov 20. PMID 29159795
- [Background] Murillo N, Valls-Sole J, Vidal J, Opisso E, Medina J, Kumru H. Focal vibration in neurorehabilitation. Eur J Phys Rehabil Med. 2014 Apr;50(2):231-42. PMID 24842220